CLINICAL TRIAL: NCT06067828
Title: A Double-Blind, Multicentre, Randomized, Three-Period, Three-Treatment, Cross-Over Study to Evaluate the Effect of BGF MDI, BFF MDI, and Placebo MDI on Exercise Parameters in Participants With COPD (ATHLOS)
Brief Title: A Study to Evaluate the Effect of Budesonide, Glycopyrronium, Formoterol Fumarate (BGF) Metered Dose Inhaler (MDI), Budesonide and Formoterol Fumarate (BFF) MDI and Placebo MDI on Exercise Parameters in Participants With Chronic Obstructive Pulmonary Disease (COPD).
Acronym: ATHLOS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D5988C00001
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Metered Dose Inhalers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BGF MDI (Active Comparator): Pressurized MDI fixed combination product of Budesonide 160 μg, Glycopyrronium 7.2 μg, and Formoterol Fumarate 4.8 μg per actuation.
  Interventions: Drug: Treatment A : Budesonide, Glycopyrronium, and Formoterol Fumarate
- BFF MDI (Active Comparator): Pressurized MDI fixed combination product of Budesonide 160 μg and Formoterol Fumarate 4.8 μg per actuation.
  Interventions: Drug: Treatment B: Budesonide and Formoterol Fumarate
- Placebo (Placebo Comparator): Placebo as pressurized inhalation suspension.
  Interventions: Drug: Treatment C : Placebo

INTERVENTIONS:
Drug: Treatment A : Budesonide, Glycopyrronium, and Formoterol Fumarate — Randomized participants will receive 2 inhalations of BGF MDI via oral inhalation twice daily (BID).
  Arms: BGF MDI
Drug: Treatment B: Budesonide and Formoterol Fumarate — Randomized participants will receive 2 inhalations of BFF MDI via oral inhalation BID.
  Arms: BFF MDI
Drug: Treatment C : Placebo — Randomized participants will receive 2 inhalations of placebo MDI via oral inhalation BID.
  Arms: Placebo

SUMMARY:
This study will investigate the effect of Budesonide, Glycopyrronium, and Formoterol Fumarate (BGF) metered dose inhaler (MDI) compared with Placebo MDI, and Budesonide and Formoterol Fumarate (BFF) MDI on isotime inspiratory capacity (IC) and exercise endurance time.

DETAILED DESCRIPTION:
This is a multicenter, three-treatment, three-period, cross-over study to assess the effect of BGF MDI vs Placebo MDI and BFF MDI in participants with COPD who have exertional breathlessness despite treatment with mono or dual COPD maintenance therapy.

Eligible participants will be randomized equally (1:1:1:1:1:1) to 1 of 6 treatment sequences. The total duration of the study for each participant will be up to 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be male or female, 40 to 80 years of age inclusive, at the time of signing the informed consent.
* Participant must have:

  * a diagnosis of COPD confirmed by a post-bronchodilator Forced expiratory volume (FEV1)/ Forced vital capacity (FVC) < 0.7 at Visit 1
  * a post-bronchodilator FEV1 ≥ 30% and <80% predicted normal (moderate to severe COPD) at Visit 1.
  * a score of ≥ 2 on the modified Medical Research Council at Visit 1.
  * pre-bronchodilator FRC of > 120% of predicted normal FRC values at Visit 1.
  * a constant work rate test endurance time of 3 to 8 minutes at Visit 2.
* Participant must be on a stable dose of mono-or dual inhaled maintenance COPD treatment for at least 6 weeks.
* Current or former smoker with a history of ≥ 10 pack-years of tobacco smoking
* Body mass index < 40 kg/m2.
* Male and Female participants (not applicable for female participants with non-childbearing potential) and their partners must use an acceptable method of contraception.

Exclusion Criteria:

* A current diagnosis of asthma, asthma- COPD-overlap, or any other chronic respiratory disease other than COPD such as alpha-1 antitrypsin deficiency, active tuberculosis, lung cancer, lung fibrosis, sarcoidosis, interstitial lung disease and pulmonary hypertension.
* Historical or current evidence of a clinically significant disease
* Participants on oxygen therapy or that desaturate significantly (<82%) during exercise.
* Participants who are enrolled or entering a pulmonary rehabilitation program during the study.
* Participants who have cancer that has not been in complete remission for at least 5 years.
* Participants with a diagnosis of narrow-angle glaucoma that has not been adequately treated and/or change in vision that may be relevant, in the opinion of the investigator.
* Participants with symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention that, in the opinion of the investigator, is clinically significant.
* Participants who have a history of hypersensitivity to β2-agonists, budesonide or any other corticosteroid components, glycopyrronium or other muscarinic anticholinergics, or any component of the MDI or dry powder inhaler.
* Participant with resting (5 minutes) oxygen saturation SaO2 in room air ≤ 85%.
* A COPD exacerbation that requires hospitalization within 12 months prior to Visit 1 or a COPD exacerbation that requires systemic corticosteroids or antibiotics within 4 months of Visit 1.
* Participants with contraindications to cardiopulmonary exercise testing (CPET).
* Participants who have had a respiratory tract infection within 8 weeks prior to Visit 1 and/or during the screening period.
* Participants with lung lobectomy, lung volume reduction or lung transplantation.
* Unable to withhold short-acting bronchodilators for 6 hours prior to lung function testing at each study visit.
* Known history of drug or alcohol abuse within 12 months.
* Any regular recreational use of marijuana in the 12 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in isotime Inspiratory capacity (IC) | 2 weeks post-treatment
  To assess the effect of BGF MDI relative to Placebo MDI and BGF MDI relative to BFF MDI on dynamic hyperinflation in participants with COPD.

SECONDARY OUTCOMES:
Change from baseline in constant work rate cycle ergometry endurance time | 2 weeks post-treatment
  To assess the effect of BGF MDI relative to Placebo MDI, BGF MDI relative to BFF MDI and BFF MDI relative to Placebo MDI on exercise endurance time in participants with COPD.
Change from baseline in Isotime dyspnea (NRS) | 2 weeks post-treatment
  To assess the effect of BGF MDI relative to Placebo MDI, BGF MDI relative to BFF MDI and BFF MDI relative to Placebo MDI on Isotime dyspnea in participants with COPD.
Change from baseline in functional residual capacity (FRC) | 2 weeks post-treatment
  To assess the effect of BGF MDI relative to BFF MDI and BFF MDI relative to Placebo MDI on FRC in participants with COPD.
Change from baseline in total lung capacity (TLC) | 2 weeks post-treatment
  To assess the effect of BGF MDI relative to BFF MDI and BFF MDI relative to Placebo MDI on TLC in participants with COPD.
Change from baseline in residual volume (RV) | 2 weeks post-treatment
  To assess the effect of BGF MDI relative to BFF MDI and BFF MDI relative to Placebo MDI on RV in participants with COPD.
Change from baseline in RV/TLC | 2 weeks post-treatment
  To assess the effect of BGF MDI relative to BFF MDI and BFF MDI relative to Placebo MDI on RV/TLC in participants with COPD.
Change from baseline in specific airway conductance (sGaw) | 2 weeks post-treatment
  To assess the effect of BGF MDI relative to BFF MDI and BFF MDI relative to Placebo MDI on sGaw in participants with COPD.
Change from baseline in static Inspiratory capacity (IC) | 2 weeks post-treatment
  To assess the effect of BGF MDI relative to BFF MDI and BFF MDI relative to Placebo MDI on static IC in participants with COPD.
Number of participants with serious adverse events (SAEs) and adverse event leading to discontinuation of study intervention (DAEs). | 2 weeks post-treatment
  To assess the safety and tolerability of BGF MDI and BFF MDI.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Tarzana, California
  - Research Site, Torrance, California
  - Research Site, Brooksville, Florida
  - Research Site, Anderson, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Spartanburg, South Carolina
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Kingston, Ontario
  - Research Site, Sainte-Foy, Quebec
- China (4):
  - Research Site, Guangzhou
  - Research Site, Nanchang
  - Research Site, Shenyang
  - Research Site, Zhengzhou
- Germany (7):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Großhansdorf
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Lübeck
  - Research Site, Mainz
- South Korea (2):
  - Research Site, Daegu
  - Research Site, Seoul
- Spain (4):
  - Research Site, Benalmádena
  - Research Site, Madrid
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- United Kingdom (3):
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/